CLINICAL TRIAL: NCT06169215
Title: A Randomized Phase 2 Study of Daratumumab-Selinexor-Velcade-Dexamethasone (Dara-SVD) for High-Risk Newly Diagnosed Multiple Myeloma
Brief Title: Comparing the Combination of Selinexor-Daratumumab-Velcade-Dexamethasone (Dara-SVD) With the Usual Treatment (Dara-RVD) for High-Risk Newly Diagnosed Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-07073; NCI-2023-07073 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10612 (Other: Yale University Cancer Center LAO); 10612 (Other: CTEP); UM1CA186689 (NIH)
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Specimen Handling; Biopsy; Bortezomib; daratumumab; Hyaluronoglucosaminidase; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Lenalidomide; Magnetic Resonance Spectroscopy; selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (Dara-SVD) (Experimental): Patients receive daratumumab and hyaluronidase-fihj SC on days 1, 8, 15, & 22 for cycles 1-2, then days 1 & 15 for cycles 3-4, and selinexor PO, bortezomib SC, and dexamethasone PO on days 1, 8, 15, & 22 of each cycle. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo PET, MRI, or CT, and bone marrow aspiration and biopsy, and collection of blood and urine samples throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Bortezomib; Procedure: Computed Tomography; Drug: Daratumumab and Recombinant Human Hyaluronidase; Drug: Dexamethasone; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Drug: Selinexor
- Arm II (Dara-RVD) (Active Comparator): Patients receive daratumumab and hyaluronidase-fihj SC on days 1, 8, 15, & 22 for cycles 1-2, then days 1 & 15 for cycles 3-4, lenalidomide PO QD on days 1-21 of each cycle, and bortezomib SC and dexamethasone PO on days 1, 8, 15, & 22 of each cycle. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo PET, MRI, or CT, and bone marrow aspiration and biopsy, and collection of blood and urine samples throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Bortezomib; Procedure: Computed Tomography; Drug: Daratumumab and Recombinant Human Hyaluronidase; Drug: Dexamethasone; Drug: Lenalidomide; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood and urine samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Bortezomib — Given SC
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; LDP-341; LDP341; MLN 341; MLN-341; MLN341; PS 341; PS-341; PS341; Velcade
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Daratumumab and Recombinant Human Hyaluronidase — Given SC
  Other Names: DARA Co-formulated with rHuPH20; DARA/rHuPH20; Daratumumab + rHuPH20; Daratumumab and Hyaluronidase; Daratumumab and Hyaluronidase-fihj; Daratumumab and vorhyaluronidase; Daratumumab and Vorhyaluronidase Alfa; Daratumumab with rHuPH20; Daratumumab-rHuPH20; Daratumumab/Hyaluronidase-fihj; Daratumumab/rHuPH20 Co-formulation; Darzalex Faspro; Darzalex/rHuPH20; Darzquro; HuMax-CD38-rHuPH20; Recombinant Human Hyaluronidase Mixed with Daratumumab
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hemady; Hexadecadrol; Hexadrol; LenaDex; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Lenalidomide — Given PO
  Other Names: CC 5013; CC-5013; CC5013; CDC 501; Revlimid
  Arms: Arm II (Dara-RVD)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Drug: Selinexor — Given PO
  Other Names: ATG-010; CRM1 Nuclear Export Inhibitor KPT-330; KPT 330; KPT-330; KPT330; Nexpovio; Selective Inhibitor of Nuclear Export KPT-330; SINE KPT-330; Xpovio
  Arms: Arm I (Dara-SVD)

SUMMARY:
This phase II trial compares the combination of selinexor, daratumumab and hyaluronidase-fihj (daratumumab), velcade (bortezomib), and dexamethasone (Dara-SVD) to the usual treatment of daratumumab, lenalidomide, bortezomib, and dexamethasone (Dara-RVD) in treating patients with high-risk newly diagnosed multiple myeloma. Selinexor is in a class of medications called selective inhibitors of nuclear export (SINE). It works by blocking a protein called CRM1, which may keep cancer cells from growing and may kill them. Daratumumab is in a class of medications called monoclonal antibodies. It binds to a protein called CD38, which is found on some types of immune cells and cancer cells, including myeloma cells. Daratumumab may block CD38 and help the immune system kill cancer cells. Bortezomib blocks several molecular pathways in a cell and may cause cancer cells to die. It is a type of proteasome inhibitor and a type of dipeptidyl boronic acid. Dexamethasone is in a class of medications called corticosteroids. It is used to reduce inflammation and lower the body's immune response to help lessen the side effects of chemotherapy drugs. Lenalidomide is in a class of medications called immunomodulatory agents. It works by helping the bone marrow to produce normal blood cells and by killing abnormal cells in the bone marrow. The drugs daratumumab, lenalidomide, bortezomib, dexamethasone and selinexor are already approved by the Food and Drug Administration for use in myeloma. But selinexor is not used until myeloma comes back (relapses) after initial treatment. Giving selinexor in the initial treatment may be a superior type of treatment for patients with high-risk newly diagnosed multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare deep response (complete response [CR] + stringent CR [sCR]) by the end of induction cycle 4 in newly diagnosed high-risk multiple myeloma patients (HR NDxMM), in both study arms.

SECONDARY OBJECTIVES:

I. To assess the minimal residual disease (MRD)-negativity (10^-5). II. To assess overall response rate (ORR), very good partial response (VGPR), and partial response (PR).

III. To assess progression-free survival (PFS) and duration of response (DOR).

CORRELATIVE OBJECTIVE:

I. To identify differential gene expression signature that predicts response to selinexor through ribonucleic acid sequencing (RNAseq) and cell-free deoxyribonucleic acid (cfDNA) studies.

EXPLORATORY THROMBOEMBOLISM RISK OBJECTIVES:

I. To estimate cumulative incidence of venous and arterial thromboembolic events.

II. To calculate IMPEDE and SAVED risk scores at baseline and at time of venous thromboembolic event.

III. To describe thromboprophylaxis strategies on treatment and venous and arterial thromboembolic events.

IV. To estimate incidence of clinically significant (major) bleeding events and assess association with thromboprophylaxis strategy.

V. To assess the association of venous and arterial thromboembolic events with PFS and all-cause mortality.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (Dara-SVD): Patients receive daratumumab and hyaluronidase-fihj subcutaneously (SC) on days 1, 8, 15, & 22 for cycles 1-2, then days 1 & 15 for cycles 3-4, and selinexor orally (PO), bortezomib SC, and dexamethasone PO on days 1, 8, 15, & 22 of each cycle. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo positron emission tomography (PET), magnetic resonance imaging (MRI), or computed tomography (CT), and bone marrow aspiration and biopsy, and collection of blood and urine samples throughout the study.

ARM II (Dara-RVD): Patients receive daratumumab and hyaluronidase-fihj SC on days 1, 8, 15, & 22 for cycles 1-2, then days 1 & 15 for cycles 3-4, lenalidomide PO once daily (QD) on days 1-21 of each cycle, and bortezomib SC and dexamethasone PO on days 1, 8, 15, & 22 of each cycle. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Treatment repeats every 28 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo PET, MRI, or CT, and bone marrow aspiration and biopsy, and collection of blood and urine samples throughout the study.

After completion of study treatment, patients are followed up at 6 months and 1 and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Presence of newly diagnosed (dx) multiple myeloma (MM) as defined by standard International Myeloma working group (IMWG).
* Presence of high risk cytogenetics using fluorescent in situ hybridization (FISH) [del(17p), t(4;14), t(14;16), t(14;20), chromosome 1 abnormalities, MYC translocation, tetrasomies, complex karyotype, high lactate dehydrogenase (LDH), or extramedullary MM.
* Patients are allowed to have received one cycle of bortezomib-based doublet or triplet therapy. For instance, if a newly diagnosed patient with MM is in need of urgent therapy, they may be enrolled after having received one cycle of bortezomib, cyclophosphamide, dexamethasone.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%).
* Absolute neutrophil count ≥ 1,000/mcL (> 500 if bone marrow [BM] clonal plasma cell involvement greater than 50%).
* Platelets ≥ 100,000/mcL (> 50,000 if BM clonal plasma cell involvement greater than 50%).
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN) (with the exception of patients with Gilbert's syndrome who have a high baseline bilirubin).
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) ≤ 3 × institutional ULN.
* Glomerular filtration rate (GFR) ≥ 30 mL/min.
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Patients with treated brain involvement are eligible if follow-up brain imaging performed within 10 days after central nervous system (CNS)-directed therapy shows no.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
* The effects of selinexor (KPT-330) on the developing human fetus are unknown. For this reason and because selective nuclear export inhibitors as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men with partners of women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men (with partners of women of childbearing potential) treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of study treatment administration. Adequate contraception should continue for 7 months for females and for 4 months for males after completion of the study treatment.
* Female of childbearing potential (FCBP) must have a negative pregnancy test during screening. They must either commit to continue abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 4 weeks before therapy, while taking lenalidomide, during dose interruptions, and for 7 months after study treatment. If menstrual cycles are irregular, the pregnancy testing should occur every 2 weeks. Pregnancy testing and counseling should be performed if a patient misses her period or if there is any abnormality in her menstrual bleeding. Lenalidomide treatment must be discontinued during this evaluation.
* Men who are sexually active with FCBP must agree to use a latex or synthetic condom while taking lenalidomide, during dose interruptions and for up to 4 weeks after discontinuing lenalidomide, even if they have undergone a successful vasectomy. Male patients taking lenalidomide must abstain from donating blood, semen, or sperm during study participation and for at least 4 weeks after discontinuation from lenalidomide.
* Patients who are randomized to receive lenalidomide need to register into the mandatory Risk Evaluation and Mitigation Strategies (REMS) program and be willing and able to comply with the requirements of REMS.
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign and give informed consent on behalf of study participants.

Exclusion Criteria:

* Patients who are in urgent need for MM therapy (such as in the setting of acute kidney injury, or high disease burden concerning for impending organ failure) may begin study treatment immediately after receiving one cycle of bortezomib combination (e.g. bortezomib-dexamethasone or cyclophosphamide-bortezomib-dexamethasone) or one course of pulse dose dexamethasone 20-40mg once daily for four days. No washout period is required.
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia.
* Patients who are receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to selinexor (KPT-330) or other agents used in study.
* Concomitant medications: Supportive care therapies such as bone directed therapies (zoledronic acid, denosumab), intravenous immunoglobulin therapy (IVIG) and anti-viral agents are allowed and recommended as per standard of care (SOC). Strong CYP3A4 inhibitors and strong CYP3A4 inducers are prohibited, due to their respective increase or decrease in bortezomib exposure. If strong CYP3A4 inhibitors cannot be avoided, then patients will be monitored for signs of bortezomib toxicity and a dose reduction of bortezomib will be considered.
* Patients with uncontrolled intercurrent illness or any other significant condition(s) that would make participation in this protocol unreasonably hazardous.
* Pregnant women are excluded because this study involves an investigational drug that may cause genotoxic, teratogenic, and mutagenic effects on the developing fetus and newborn and drugs that have known genotoxic, teratogenic, or abortifacient effect.

  * Because there is potential risk for adverse events in nursing infants secondary to treatment of the mother with the drugs used in this study, breastfeeding is not allowed during treatment for all drugs and for 2 months after last dose of bortezomib and 1 week after the last dose of selinexor.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Deep clinical response | Up to the end of cycle 4 (each cycle = 28 days)
  Defined as complete response (CR) + stringent CR.

SECONDARY OUTCOMES:
Minimal residual disease-negativity (10^-5) | Up to end of cycle 4 (each cycle = 28 days)
  Will be assessed by next generation flow cytometry.

OTHER OUTCOMES:
Ribonucleic acid (RNA) and cell free deoxyribonucleic acid (DNA) sequencing | Baseline up to end of cycle 4 (each cycle = 28 days)
  Will compare pre- and post-treatment RNA and cell free DNA sequencing data to identify unique differential signature correlated with deep responses among subjects treated with selinexor-daratumumab-velcade-dexamethasone regimen. Will use cox proportional hazard models to identify a gene signature predictive of response to selinexor.
Venous thromboembolism | Up to 2 years
  Venous thromboembolism will be a composite endpoint comprised of adverse events associated with study medications defined according to Common Terminology Criteria for Adverse Events grade, term and system organ class as follows: grades 1-5 thromboembolic events; grades 2-5 portal vein thrombosis; grades 1-5 superior vena cava syndrome; grades 1-5 vascular access complication; grades 3-5 arterial thromboembolism.
Incidence of adverse events associated with anticoagulation thromboprophylaxis strategy | Up to 2 years
  Will be defined as follows: clinically significant major bleeding events including required transfusion of red blood cells; required admission to the hospital for > 24 hours; prolonged hospitalization, with bleeding as the principal reason; required surgery to stop the bleeding.
Venous thromboembolism risk factors | At baseline and at the time of incidence of venous thromboembolism
  All the data comprising two established risk scores, IMPEDE or SAVED, will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Neparidze, Principal Investigator — Yale University Cancer Center LAO
Locations (27):
- United States (27):
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UCI Health Laguna Hills, Laguna Hills, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - NYU Langone Hospital - Brooklyn, Brooklyn, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm